CLINICAL TRIAL: NCT03361774
Title: A Clinical Method Development Study to Characterise The Efficacy of An Experimental Dual Active Combination Dentifrice For The Relief Of Dentin Hypersensitivity
Brief Title: A Clinical Method Development Study to Characterise The Efficacy of a Dentifrice For The Relief Of Dentin Hypersensitivity
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Cancelled before Active
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 208675
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical examiner will be blinded to treatment received. The study statistician, data management staff, other employees of the Sponsor and vendors acting on behalf of the sponsor, who may influence study outcomes will also be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test dentifrice (Experimental): Participants in this arm will receive experimental dentifrice containing 5% w/w KNO3 and 0.454% w/w SnF2 (1100 parts per million [ppm] fluoride).
  Interventions: Drug: Dentifrice containing 5% w/w KNO3 and 0.454% w/w SnF2 (1100 ppm fluoride).
- Control dentifrice (Active Comparator): Participants in this arm will receive comparator dentifrice containing 0.454% SnF2 (1100ppm fluoride).
  Interventions: Drug: Dentifrice containing 0.454% w/w SnF2 (1100 ppm fluoride).

INTERVENTIONS:
Drug: Dentifrice containing 5% w/w KNO3 and 0.454% w/w SnF2 (1100 ppm fluoride). — Participants will be instructed to dose the toothbrush with a strip of dentifrice containing 5% w/w KNO3 and 0.454% w/w SnF2 (1100 ppm fluoride) (a full brush head) and brush for at least 1 timed minute, twice daily (morning and evening), making sure to brush all sensitive areas of their teeth.
  Participants will be permitted to rinse with tap water post-brushing if they wish to.
  Arms: Test dentifrice
Drug: Dentifrice containing 0.454% w/w SnF2 (1100 ppm fluoride). — Participants will be instructed to dose the toothbrush with a strip of dentifrice containing 0.454% w/w SnF2 (1100 ppm fluoride) (a full brush head) and brush for at least 1 timed minute, twice daily (morning and evening), making sure to brush all sensitive areas of their teeth. Participants will be permitted to rinse with tap water post-brushing if they wish to.
  Arms: Control dentifrice

SUMMARY:
The aim of this study is to develop the clinical methodology to characterize the efficacy profiles of an experimental 5% potassium nitrate (KNO3) and 0.454% stannous fluoride (SnF2) combination dentifrice and a marketed desensitizing 0.454% SnF2 only dentifrice for the relief of dentin hypersensitivity (DH), at multiple time points, over an 8 week treatment period.

DETAILED DESCRIPTION:
This will be a single center, 8 week, randomized, controlled, examiner blind, two treatment arm, parallel design, stratified (by maximum baseline Schiff sensitivity score of the two selected test teeth), method development study, in participants in good general health, with pre-existing self-reported tooth sensitivity, and at least two sensitive teeth (diagnosed clinically) that meet all study criteria at the screening and baseline (pre-treatment) visits.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent form (ICF) indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee: a) No clinically significant and relevant abnormalities in medical history or upon oral examination. b) Absence of any condition that would impact the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.
* Male participant able to father children, or female participant of child-bearing potential and at risk for pregnancy, must agree to use a highly effective method of contraception throughout the study and for at least 5 days after the last dose of assigned treatment. Female participant not of child-bearing potential must meet requirements as follows: Achieved post-menopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months, with no alternative pathological or physiological cause, and have a serum follicle-stimulating hormone (FSH) level confirming post-menopausal state, Have undergone a documented hysterectomy and/or bilateral oophorectomy, Have medically confirmed ovarian failure.
* AT Visit 1 (Screening): participant must have a) Self-reported history of DH lasting more than six months but not more than 10 years. b) Minimum of 20 natural teeth. c) Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria: Signs of facial/cervical erosion, abrasion or gingival recession (EAR), Tooth with MGI score = 0 adjacent to the test area (exposed dentin) only and a clinical mobility of ≤1, Tooth with signs of sensitivity, as evidenced by qualifying tactile (tactile threshold ≤ 20g) and evaporative air (Schiff sensitivity score ≥ 2) sensitivity.
* AT Visit 2 (Baseline): participant must have a minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), preferably in different quadrants, with signs of sensitivity, as evidenced by qualifying tactile (tactile threshold ≤ 20g) and evaporative air (Schiff sensitivity score ≥ 2) sensitivity at both Screening and Baseline. All teeth which meet the sensitivity criteria (tactile threshold ≤ 20g; Schiff sensitivity score ≥ 2) at Screening (Visit 1) should be assessed by tactile stimulus at Baseline (Visit 2). Those teeth which meet the required tactile threshold (Yeaple ≤20g) again at Baseline should then be assessed by evaporative air stimulus. The examiner will select two 'Test Teeth' from those which meet the tactile threshold and Schiff sensitivity score inclusion criteria at Screening and Baseline. Once these two teeth have been identified, no further testing is necessary. Test Teeth should not be adjacent to each other and preferably in different quadrants.

Exclusion Criteria:

* An employee of the investigational site directly involved in the conduct of the study or a member of their immediate family; an employee of the investigational site otherwise supervised by the investigator; a GSK employee directly involved in the conduct of the study or a member of their immediate family.
* Participation in other studies (including cosmetic studies) involving investigational drug(s) within 30 days of study entry and/or during study participation.
* Participation in another tooth desensitizing treatment study within 8 weeks Screening.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Pregnant female participant (as evidenced by a positive urine pregnancy test).
* Breastfeeding female participant.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Recent history (within the last year) of alcohol or other substance abuse.
* Dental prophylaxis within 4 weeks of Screening.
* Tongue or lip piercing or presence of multiple dental implants.
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Participant with evidence of gross intra-oral neglect or the need for extensive dental therapy.
* Teeth bleaching within 8 weeks of Screening.
* Participant with fixed or removable partial dentures.
* Participant with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.
* Specific exclusions for test teeth: a) Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening, b) Tooth with exposed dentin but with deep, defective or facial restorations, c) Teeth with full crowns or veneers, d) Sensitive teeth with contributing etiologies other than erosion, abrasion or recession of exposed dentin, e) Sensitive tooth not expected to respond to treatment with an over-the-counter dentifrice in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentin hypersensitivity within 8 weeks of Screening (participant will be required to bring their current oral care products to the site in order to verify the absence of known anti-sensitivity ingredients).
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, anti-depressants, mood-altering and anti-inflammatory drugs.
* Use of antibiotics in the 2 weeks prior to the Screening visit, or in the 2 weeks prior to the Baseline visit during the acclimatization period.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia.
* Participant who requires antibiotic prophylaxis for dental procedures.
* Participant who is unwilling or unable to comply with the Lifestyle/Study Restrictions described in the study protocol.
* Participant who has previously been enrolled in this study.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2018-12-03 (Estimated); Study Completion 2018-12-03 (Estimated)

PRIMARY OUTCOMES:
Mean Schiff Sensitivity Score at Baseline (Day 0) | Baseline (Day 0)
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the selected two test teeth at baseline.
Mean Schiff Sensitivity Score at Day 3 | Day 3
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the two test teeth on Day 3.
Mean Schiff Sensitivity Score at Day 7 | Day 7
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the two test teeth on Day 7.
Mean Schiff Sensitivity Score at Day 14 | Day 14
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the two test teeth on Day 14.
Mean Schiff Sensitivity Score at Day 28 | Day 28
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the two test teeth on Day 28.
Mean Schiff Sensitivity Score at Day 56 | Day 56
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. Lesser the Schiff sensitivity score, lesser is the sensitivity of the tooth. Mean score will be calculated as the average score of the two test teeth on Day 56.
Mean Tactile Threshold at Baseline (Day 0) | Baseline (Day 0)
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Baseline (Day 0).
Mean Tactile Threshold at Day 3 | Day 3
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Day 3.
Mean Tactile Threshold at Day 7 | Day 7
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Day 7.
Mean Tactile Threshold at Day 14 | Day 14
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Day 14.
Mean Tactile Threshold at Day 28 | Day 28
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Day 28.
Mean Tactile Threshold at Day 56 | Day 56
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g. Mean score will be calculated as the average score of the two test teeth on Day 56.
Change From Baseline (Day 0) in Schiff Sensitivity Score on Day 3 | Baseline (Day 0), Day 3
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score will indicate the improvement in sensitivity.
Change From Baseline (Day 0) in Schiff Sensitivity Score on Day 7 | Baseline (Day 0), Day 7
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score will indicate the improvement in sensitivity.
Change From Baseline (Day 0) in Schiff Sensitivity Score on Day 14 | Baseline (Day 0), Day 14
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score will indicate the improvement in sensitivity.
Change From Baseline (Day 0) in Schiff Sensitivity Score on Day 28 | Baseline (Day 0), Day 28
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score will indicate the improvement in sensitivity.
Change From Baseline (Day 0) in Schiff Sensitivity Score on Day 56 | Baseline (Day 0), Day 56
  The examiner will assess the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale scored as follows - 0: Participant does not respond to air stimulation; 1: responds to air stimulus but does not request discontinuation of stimulus; 2: Participant responds to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. A reduction in Schiff Sensitivity score will indicate the improvement in sensitivity.
Change From Baseline (Day 0) in Tactile Threshold on Day 3 | Baseline (Day 0), Day 3
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g.
Change From Baseline (Day 0) in Tactile Threshold on Day 7 | Baseline (Day 0), Day 7
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g.
Change From Baseline (Day 0) in Tactile Threshold on Day 14 | Baseline (Day 0), Day 14
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g.
Change From Baseline (Day 0) in Tactile Threshold on Day 28 | Baseline (Day 0), Day 28
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g.
Change From Baseline (Day 0) in Tactile Threshold on Day 56 | Baseline (Day 0), Day 56
  The examiner will assess the response to tactile sensitivity using a Yeaple probe which will allow application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force will reach. The tactile threshold for each tooth will be determined by asking the participants whether the sensation caused discomfort. The pressure setting at which the participant will give two consecutive 'yes' responses will be recorded as the tactile threshold. Higher tactile threshold will indicate the less sensitive are the tooth. At baseline, the maximum force will be 20g; at all subsequent visits, it will be 80g. However, in situations where participants will not give a 'yes' response at force of 80g, the tactile threshold will be recorded as >80g.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 0 (Baseline) | Baseline (Day 0)
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 3 | Day 3
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 7 | Day 7
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 14 | Day 14
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 28 | Day 28
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Number of sensitive teeth (Schiff sensitivity score ≥ 1) on Day 56 | Day 56
  The number of teeth with a Schiff sensitivity score of ≥1 will be consider sensitive teeth. Schiff sensitivity scores were as follows:0= Subject does not respond to air stimulation, 1= if participants respond to air stimulus but does not request discontinuation of stimulus; 2= participants respond to air stimulus and requests discontinuation or moves from stimulus; 3 = participants respond to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: No